CLINICAL TRIAL: NCT01929083
Title: Influence of Progesterone Administration on Drug-Induced QT Interval Prolongation and Torsades de Pointes
Brief Title: Influence of Progesterone Administration on Drug-Induced QT Interval Lengthening
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, James E. Tisdale, Professor of Pharmacy Practice, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12GRNT12060187
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Results first posted 2015-09-28 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Prolonged QT Interval in EKG and Sudden Death
Keywords: Torsades de pointes; Progesterone; Clinical trial; Risk reduction; Electrocardiography
MeSH Terms: conditions — Jervell-Lange Nielsen Syndrome; Torsades de Pointes; Risk Reduction Behavior | interventions — Progesterone; ibutilide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Experimental): Subjects will receive treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days
  Interventions: Drug: Progesterone; Drug: Ibutilide
- Placebo (Placebo Comparator): Subjects will receive oral placebo, two capsules once daily every evening for 7 days
  Interventions: Drug: Placebo; Drug: Ibutilide

INTERVENTIONS:
Drug: Progesterone — Subjects will receive oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
  Arms: Progesterone
Drug: Placebo — Subjects will receive oral placebo two capsules once daily every evening for 7 days
  Arms: Placebo
Drug: Ibutilide — Ibutilide 0.003 mg/kg administered to all subjects to moderately lengthen the QT interval

SUMMARY:
Female sex is an independent risk factor for the potentially fatal drug-induced arrhythmia (irregular heartbeat) known as torsades de pointes (TdP), which is associated with prolongation of the corrected QT (QTc) interval on the electrocardiogram (ECG). Mechanisms for this increased risk in women are not well-understood. QTc interval duration has been shown to fluctuate throughout the phases of the menstrual cycle. Evidence indicates that the QTc interval response to drugs that may cause TdP is greater during the menses and ovulation phases of the menstrual cycle, during which serum progesterone concentrations are lowest, and lesser during the luteal phase, during which serum progesterone concentrations are highest. Additional evidence from our laboratory suggests that progesterone may be protective against TdP. Specific Aim 1: Establish the influence of oral progesterone administration as a preventive method by which to diminish the degree of drug-induced QT interval prolongation in women. Working hypothesis: Oral progesterone administration effectively attenuates enhanced drug-induced QT interval response in women. To test this hypothesis, progesterone or placebo will be administered in a crossover fashion to women during the menses phase of the menstrual cycle. QTc interval response to low-dose ibutilide, a drug known to lengthen the QT interval, will be assessed. The primary endpoint will be individually-corrected QT interval (QTcI) response to ibutilide, in the presence and absence of progesterone, which will be assessed by: 1) Effect on maximum change in QTcI, and 2) Area under the QTcI interval-time curves (AUEC). At the conclusion of this study, we will have established that oral progesterone administration is a safe and effective method of attenuating drug-induced QT interval prolongation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 21-40 years
* Premenopausal

Exclusion Criteria:

Serum potassium ,< 3.6 meq/l

* Serum magnesium < 1.8 mg/dl
* Serum hemoglobin < 9.0 mg/dl
* Serum hematocrit < 26%
* Hypertension
* Coronary artery disease
* Heart failure
* Liver disease
* Kidney disease
* Serum creatinine > 1.5 mg/dl
* Taking hormone contraceptives
* Baseline Bazett's correct QTc interval > 450 ms
* Family history of long-QT syndrome, arrhythmias, sudden cardiac death
* Concomitant use of any QT prolonging drug
* Pregnancy
* weight < 45 kg
* Unwillingness to use non-hormonal forms of birth control during the study period

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Tisdale, BSc, PharmD, Principal Investigator — Purdue University & Indiana University
Locations (2):
- United States (2):
  - Indiana Clinical Research Center, Indianapolis, Indiana
  - Purdue University, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from a) INResearch database, maintained by Indiana Clinical Translational Research Institute (CTSI), and b) Hard copy and electronic advertisements on the IUPUI and Purdue University campuses Participants were recruited between October 2012 and February 2014
Pre-assignment Details: n=333 subjects assessed for eligibility; n=27 consented, n=306 excluded (n=108 did not meet inclusion criteria, n=198 declined to participate); of n=27 consented, n=19 enrolled, n=8 excluded because they met one or more exclusion criteria
Groups:
- Progesterone First, Then Placebo: Subjects will receive treatment with oral progesterone 400 mg once daily (two x 200 mg capsules) every evening for 7 days
  Progesterone: Subjects will receive oral progesterone 400 mg (two x 200 mg capsules) once daily every evening for 7 days
- Placebo First, Then Progesterone: Subjects will receive oral placebo, two capsules once daily every evening for 7 days
  Placebo: Subjects will receive oral placebo two capsules once daily every evening for 7 days
Period: Intervention 1
Arm/Group | Progesterone First, Then Placebo | Placebo First, Then Progesterone
Started | 10 (Number of patients randomized to receive progesterone first) | 9
Returned for 1st Ibutilide Administratio | 7 | 9
Completed | 7 | 9
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Nonadherent to study medications | 1 | 0
Period: Intervention 2
Arm/Group | Progesterone First, Then Placebo | Placebo First, Then Progesterone
Started | 7 | 9
Returned for 2nd Ibutilide Administratio | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Includes n=15 subjects included in the final analysis. Includes subjects randomized to receive progesterone first and patients randomized to receive placebo first
Groups:
- Entire Study Population: n=15 subjects who completed the study
Arm/Group | Entire Study Population
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Baseline (Pre-Ibutilide) QTcI Intervals
Time Frame: After 7 days of progesterone or placebo, prior to receiving IV ibutilide
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 15 | 15
ms | 412 (15) | 419 (14)
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.04, t-test, 2 sided; Paired t-test

2. Primary Outcome: Maximum Individual-corrected QT Interval (QTcI)
Description: QT intervals will be corrected as follows: Prior to randomization, subjects will come to the Indiana Clinical Research Center for a 12-hour stay, during which three ECGs, one minute apart, will be obtained at the following times: 0, 15 & 30 minutes, and 1, 2, 4, 6, 8, and 12 hours. Subjects will be discharged, and then return then next morning for the 24 hour ECG. QT and RR intervals will be used to determine each subject's individual rate-corrected QT interval (QTcI) using the parabolic model QT = β•RRα, where RR is the interval between adjacent QRS complexes, and α and β are subject-specific correction factors.
Time Frame: 0, 15 & 30 minutes, and 1, 2, 4, 6, 8, and 12 hours post-ibutilide administration
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 15 | 15
ms | 443 (17) | 458 (19)
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.003, t-test, 2 sided; Paired t-test

3. Secondary Outcome: Incidence of Progesterone-associated Adverse Effects Compared to Placebo
Time Frame: During 7 days of treatment with oral progesterone or placebo
Measure: Number; unit: percentage of participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 16 | 17
percentage of participants
  Fatigue/general malaise | 38 | 6
  Headache | 13 | 6
  Mood changes | 13 | 0
  Breast tenderness | 13 | 0
  Hypotension | 6 | 0
  Vertigo requiring discontinuation | 6 | 0
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.04, Fisher Exact — P value for incidence of fatigue/malaise
Statistical Analysis 2: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.60, Fisher Exact — p values for incidence of headache
Statistical Analysis 3: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.23, Fisher Exact — p value for incidence of mood changes
Statistical Analysis 4: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.23, Fisher Exact — p value for incidence of breast tenderness
Statistical Analysis 5: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.48, Fisher Exact — p value for incidence of hypotension
Statistical Analysis 6: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.48, Fisher Exact — p value for incidence of vertigo requiring discontinuation of therapy

4. Primary Outcome: Maximum % Change From Baseline in QTcI Intervals Following Ibutilide Administration
Time Frame: After 7 days of progesterone or placebo
Measure: Mean (Standard Deviation); unit: percentage change from baseline value
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 15 | 15
percentage change from baseline value | 7.5 (2.4) | 9.3 (3.4)
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.02, t-test, 2 sided; Paired t-test

5. Primary Outcome: Area Under the QTcI - Time Curve (AUEC)
Time Frame: From beginning of 10-minute ibutilide infusion to 1 hour following ibutilide infusion
Measure: Mean (Standard Deviation); unit: ms*hr
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 15 | 15
ms*hr | 497 (13) | 510 (16)
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided; Paired t-test

6. Other Pre Specified Outcome: Adverse Effects Associated With Ibutilide in the Progesterone and Placebo Phases
Time Frame: Within 8 hours following ibutilide administration
Measure: Number; unit: percentage of participants
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 15 | 17
percentage of participants
  Bradycardia (HR < 60 bpm) | 20 | 12
  Burning at infusion site | 7 | 6
  Transient QTc interval > 500 ms | 0 | 6
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.65, Fisher Exact — p value for bradycardia
Statistical Analysis 2: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p > 0.99, Fisher Exact — p value for burning at infusion site
Statistical Analysis 3: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p > 0.99, Fisher Exact — p value for transient QTc interval > 500 ms

7. Other Pre Specified Outcome: Maximum (Peak) Serum Ibutilide Concentrations During Progesterone and Placebo Phases
Time Frame: Within 1 hour following ibutilide administration (0, 15 & 30 minutes and 1 hours.)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 15 | 15
pg/mL | 1247 (770) | 1172 (709)
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.43, t-test, 2 sided; Paired t-test

8. Other Pre Specified Outcome: Serum Estradiol Concentrations During the Progesterone and Placebo Phases
Time Frame: Following 7 days of progesterone or placebo
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 15 | 15
pg/mL | 89.3 (62.8) | 71.8 (31.7)
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.36, t-test, 2 sided; Paired t-test

9. Other Pre Specified Outcome: Serum Progesterone Concentrations During Progesterone and Placebo Phases
Time Frame: After 7 days of progesterone or placebo
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 15 | 15
ng/mL | 16.2 (11.0) | 1.2 (1.0)
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Paired t-test

10. Other Pre Specified Outcome: Ratio of Serum Progesterone:Estradiol Concentrations During the Progesterone and Placebo Phases
Time Frame: After 7 days of progesterone or placebo
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 15 | 15
Ratio | 205 (40) | 18 (16)
Statistical Analysis 1: Comparison: Progesterone vs Placebo; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided; Paired t-test

ADVERSE EVENTS:
Time Frame: During 7 days of therapy with progesterone or placebo
Arm/Group | Progesterone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/17
Other Adverse Events (participants affected / at risk) | 9/16 | 2/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone (N=16) | Placebo (N=17)
Vertigo requiring discontinuation of therapy (Ear and labyrinth disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone (N=16) | Placebo (N=17)
Fatigue/general malaise (General disorders) | 6 (6) | 1 (1)
Headache (General disorders) | 2 (2) | 1 (1)
Mood changes (General disorders) | 2 (2) | 0 (0)
Breast tenderness (Endocrine disorders) | 2 (2) | 0 (0)
Hypotension (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes